CLINICAL TRIAL: NCT04953455
Title: Translation and Verification of English Lysholm Knee Scoring Scale
Status: Completed | Type: Observational
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: M2016001
Record Dates: First submitted 2021-06-28; First posted 2021-07-08 (Actual); Last update posted 2021-07-08 (Actual); Status verified 2021-07

CONDITIONS: Evaluations, Diagnostic Self

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (4):
- pre-operation: Within one month before operation of diagnoses with a ligament rupture, patella dislocation, meniscus injury, or total knee replacement surgery
  Interventions: Other: no intervention
- early after operation: Within three months after operation of ligament rupture, patella dislocation, meniscus injury, or total knee replacement surgery
  Interventions: Other: no intervention
- lately after operation: within three months to one year after operation of ligament rupture, patella dislocation, meniscus injury, or total knee replacement
  Interventions: Other: no intervention
- healthy volunteers: Healthy people without abnormalities
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Through the translation and verification of the Lysholm Knee Score Scale, a Chinese version of the Lysholm Knee Score Scale supported by experimental data was obtained. And on this basis, explore the knee joint score scale that fits the Chinese situation

DETAILED DESCRIPTION:
Lysholm Knee Scoring Scale needs to be translated and back translated into Chinese version of Lysholm Knee Scoring Scale. Through data collection and analysis, the reliability, validity and sensitivity of the Chinese version of the Lysholm Knee Score Scale were studied, and on this basis, the advantages and disadvantages of the scale were analyzed, and a new knee score scale was developed based on the domestic situation.

ELIGIBILITY:
Inclusion Criteria:

* Patients with ruptured ligaments, dislocation of the patella, meniscus injury or total knee replacement before and after surgery, and have the ability to read or communicate with others normally.

Exclusion Criteria:

* Patients with other injuries to the joints of the lower limbs, or patients who do not have the ability to read or communicate with others normally.

Ages: 18 Years to 80 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Through the diagnosis of MRI and clinicians, patients who are determined to be ligament rupture, patella dislocation, meniscus injury or total knee replacement surgery before and after surgery, the patient should have the ability to read or communicate with others normally, and the age range is 18-80 years old .
Sampling Method: Non-Probability Sample
Enrollment: 92 (Actual)
Dates: Start 2017-04-01 (Actual); Primary Completion 2017-04-11 (Actual); Study Completion 2017-09-30 (Actual)

PRIMARY OUTCOMES:
Chinese version of Lysholm Knee Score Scale | 1 year after operation
  Chinese version of Lysholm Knee Score Scale
IKDC Knee Joint Score Scale | 1 year after operation
  IKDC Knee Joint Score Scale

CONTACTS AND LOCATIONS:
Overall Officials: yingfang ao, M.D., Study Chair — Peking University Third Hospital
Locations (1):
- Peking university third hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided